CLINICAL TRIAL: NCT04875611
Title: Phase II Study Evaluating the Efficacy of Nivolumab in the Treatment of Patients With Nasopharyngeal Cancer Who Progressed During or After Platinum-based Chemotherapy
Brief Title: Nivolumab in Nasopharyngeal Cancer With Progression During or After Platinum-based Treatment
Acronym: NIVONASO-21
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-NIO-0003
Record Dates: First submitted 2021-04-25; First posted 2021-05-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental therapy:OPDIVO (Nivolumab) (Experimental)
  Interventions: Drug: Opdivo

INTERVENTIONS:
Drug: Opdivo — Dose of Nivolumab is constant and is 240 mg .All patients will undergo maximum of 12 cycles of investigation product's infusion ( around 6 month of treatment).Each cycle will be done in intervals of 14 day (no less than 12 days after previous infusion and no longer than 42 day/6 weeks after previous infusion).
  Other Names: Nivolumab

SUMMARY:
Multicentre , non-randomized, prospective clinical trial to assess efficacy of Nivolumab in treatment of nasopharyngeal cancer who progressed during or after platinum-based chemotherapy . Patients disqualified from radical therapy . The total number of patients was estimated for 32.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Histological or cytological documentation of squamous cell carcinoma.
3. Primary tumor location in nasopharynx
4. Previous, documented failure on platinum-based chemotherapy or progression of the disease during platinum-based chemotherapy
5. Tumor recurrence (local or nodal) or generalization (metastasis) occurence during or within 6 months after previous platinum-based chemotherapy
6. ECOG(Eastern Cooperative Oncology Group) performance scale 0-1
7. Participant is willing and able to give informed consent for participation in the study and agrees to undergo all follow up visit and planned procedures.

Exclusion Criteria:

1. Known active central nervous system metastases.
2. Presence of renal insufficiency defined as eGFR(estimated glomerular filtration rate) < 30 ml/min/m2
3. Presence of liver disfunction, defined as level of AST(aspartate aminotransferase) and /or ALT(alanine aminotransferase) > 2,5 x ULN(upper limits of normal) (> 5 x ULN in patients with documented liver metastases); total bilirubin > 1,5 xULN ( bilirubin > 1,5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%) or albumin < 2,5 g/dL
4. Abnormalities in blood count such as: hemoglobin < 9 g/dl, platelets < 100 x 109 /L, Absolute Neutrophil Count (ANC) <1,0 x 109 /L
5. Ejection fraction in echocardiography < 50%
6. History of active autoimmune diseases except for type I diabetes, hypothyroidism (treated only with hormone supplementation), psoriasis, albinism.
7. Patient with diagnosed mental disorder preventing, in Investigator's opinion, from participating in a clinical trial.
8. Pregnancy or breastfeeding.
9. Female with childbearing potential or male participant with female partner of childbearing potential, who is unwilling or unable to use an acceptable method of contraception to avoid pregnancy throughout the entire clinical trial period and for 5 months after the end of treatment (last infusion)
10. Prior therapy with an anti-PD-1/L1/L2 and/or anti-ICOS directed agent
11. Patient is currently participating in another clinical trial.
12. Active infection, which significantly affects the patient's clinical condition and requires treatment.
13. Patient with prior bone marrow or solid organ transplantation.
14. Patient requires immunosuppressive agents, including steroids (daily dose of prednisone or equivalent > 10 mg)
15. Known immunodeficiency including HIV/AIDS(human immunodeficiency virus/acquired immunodeficiency syndrome) infection.
16. Patient received any live vaccine within 28 days before enrollment.
17. Heart Failure - NYHA(New York Heart Association functional classification system) III or IV
18. Coexistence of active malignant tumor or history of malignant tumor after radical treatment with disease-free period > 2 years, except: cervical cancer in situ/ basocellular skin cancer/prostate cancer, after radical treatment.
19. Other comorbidities symptoms or conditions that in Investigator's judgement prevent patient from participation in clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 weeks
  Percentage of objective responses (partial and complete responses combined /partial response (PR)+ complete response(CR)/ by immune Response Evaluation Criteria in Solid Tumours (iRECIST) response criteria) in MRI (Magnetic Resonance Imaging) after 12 weeks.
  1. Partial response - at least a 30% decrease in the sum of the LD(longest diameter) of target lesions, taking as reference the baseline sum LD(longest diameter)
  2. Complete response (CR)- disappearance of all target lesions and short dimension of all lymph nodes < 10 mm

SECONDARY OUTCOMES:
1.Progression- free survival (PFS) by iRECIST( immune Response Evaluation Criteria in Solid Tumours) criteria- from the beginning of treatment to the progression of disease or death. | 6 month of treatment phase
  Progression will be evaluated in MRI(Magnetic Resonance Imaging) and defined according to iRECIST(immune Response Evaluation Criteria in Solid Tumours) criteria:
  * least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) and the sum must also demonstrate an absolute increase of at least 5 mm.
  * the appearance of one or more new lesions
Overall survival (OS) rate- time of total survival | at 6 months (treatment phase), 12 months and 18 months (6th month and 12th month of long term follow up)
DCR(disease control rate) per RECIST (Response Evaluation Criteria in Solid Tumours) | through study completion, an average of 6 months
  Defined as not meeting the criteria for progression and PR(partial response)
DoR(duration of response) per RECIST (Response Evaluation Criteria in Solid Tumours) | through study completion, an average of 1 year
  Measured in MRI(Magnetic Resonance Imaging) from the time when measurement criteria for complete/ partial response are met till time when progression of the disease is documented.
Change in quality of life in EORTC QLQ-C30(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) (version 3.0) .A high scale score represents a higher response level. | from first infusion to last follow up ( 3 month, 6 month, 9 month,12month follow up)
Safety assessment of treatment with Nivolumab measured by excesive toxity | Each visit during treatment phase -12 cycles of investigation product's infusion (around 6 month of treatment).

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Klinika Hematologii z Pododziałem Chorób Naczyń Uniwersyteckiego Szpitala Klinicznego w Białymstoku, Bialystok
  - Klinika Hematologii i Transplantologii Gdańskiego Uniwersytetu Medycznego, Gdansk
  - Klinika Transplantacji Szpiku i Onkohematologii Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy, Oddział w Gliwicach, Gliwice
  - Klinika Hematologii i Transplantacji Szpiku, Świętokrzyskie Centrum Onkologii, Kielce